CLINICAL TRIAL: NCT04393987
Title: Effect Of Treatment Compliance Training Given To Patients With Bipolar Disorder On Treatment Compliance, Social Functioning, And Quality Of Life
Brief Title: Effect Of Treatment Compliance Training Given To Patients With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, ebru başkaya, Principal Investigator, Uşak University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ebaskaya
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Quality of Life; Treatment Compliance
Keywords: bipolar disorder; Treatment Compliance Training; Quality of Life; Social Functioning
MeSH Terms: conditions — Patient Compliance; Bipolar Disorder; Social Adjustment

STUDY DESIGN:
Intervention Model Description: The research was using quasi-experimentally research methods. The research was carried out with 19 patients enrolled in the Community Mental Health Center and 21 outpatients who were monitored in the Psychiatry Outpatient Clinic of a university and who met the inclusion criteria. The data were collected using the Participant Information Form, Medication Adherence Rating Scale, Social Functioning Scale, and World Health Organization Quality of Life Instrument Short Form. Treatment compliance training was given to the intervention group (n=19) individually once a week for a total of five sessions. No intervention was applied to the control group (n=21) following the pretest application. Post-tests were applied to the intervention group after the training and follow-up tests were applied to both groups three months after the training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arms (Experimental): Treatment Compliance Training The treatment compliance training consists of five sessions in total and was given individually. Each session of the treatment compliance training given once a week took 45 minutes on average.
  Interventions: Behavioral: Treatment Compliance Training
- Control Group (No Intervention): No intervention was performed on the patients in the control group, and routine follow-up (arranging treatment by the doctor, answering the patient's and family's questions about treatment) continued in the polyclinic.

INTERVENTIONS:
Behavioral: Treatment Compliance Training — Treatment Compliance Training consist of: Introduction of Treatment Compliance Program and Information about the Disease, Therapies for Bipolar Disorder and Importance of Treatment Compliance, Drugs Used for Bipolar Disorder, Effects and Side effects, Strategies to Solve Treatment-Related Problems and Cope with Stress, Beliefs, Attitudes, and Stigmatization Towards Patient/Disease in Bipolar Disorder. The sessions were held in the form of PowerPoint presentations. In the Treatment Compliance Training, lecture, question-answer, homework, sharing experiences, video presentation, summarization were used.The day before each session, patients were phoned and reminded of the time of the session.
  Arms: Arms

SUMMARY:
In bipolar disorder, treatment noncompliance is associated with high rates of recurrence and hospitalization. Furthermore, it is reported that that treatment noncompliance disturbs the social functioning of patients and reduces the quality of life. Improvement of the quality of life, social functioning and treatment compliance is as important as the long-term treatment of symptoms.This study aimed to determine the effect of treatment compliance training given to patients with bipolar disorder on treatment compliance, social functioning, and quality of life.

DETAILED DESCRIPTION:
The aim is to determine the effect of treatment compliance training given to patients with bipolar disorder on treatment compliance, social functioning, and quality of life.

The study was conducted with 38 bipolar disorder (n=17 intervention group; n=21 control group) using a quasi-experimental research design. Patients were evaluated using a pre-test, post-test, monitoring test, "Medication

Adherence Rating Scale (MARS)", "Social Functioning Scale (SFS)", and "World Health Organization Quality of Life Instrument Short Form (WHOQOLBREF-TR)." The measurements were taken 3 times:

pre test, post-test and 3-months post-test.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate,
* Being diagnosed with bipolar disorder,
* Being in the euthymic period,
* Being at the age of 18 or over,
* Being literate.

Exclusion Criteria:

* Being in an acute period of exacerbation
* Actively using alcohol or psychoactive substances
* Having another psychiatric illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Medication Adherence Rating Scale (MARS) | Change from baseline to 5 weeks (also assessed at 17 weeks post-baseline)
  The scale assesses the patient's compliance behaviors and attitude to treatment. The scale consists of 10 questions to answer in the form of Yes/No (between 1-7 were poor in compliance with treatment and those with scores between 8-10 were high). The scale assesses the patient's compliance behaviors and attitude to treatment. The scale consists of 10 questions to answer in the form of Yes/No (between 1-7 were poor in compliance with treatment and those with scores between 8-10 were high).
Social Functioning Scale (SFS) | Change from baseline to 5 weeks (also assessed at 17 weeks post-baseline)
  The Social Functioning Scale is a tool that evaluates role functions requiring judgment on the social role of an individual. The scale consists of seven subscales. The total score that can be obtained from this scale ranges between 0-223 points. High scores taken from each subscale indicate that there is a positive development in functioning.
World Health Organization Quality of Life Instrument Short Form (WHOQOLBREF-TR) | Change from baseline to 5 weeks (also assessed at 17 weeks post-baseline)
  World Health Organization Quality of Life Instrument Short Form consists of 26 questions and four domains. These 4 domains are physical health, psychological health, social relationships, and environment.Domain I: Physical domain: It covers the ability to conduct daily tasks, commitment to medicines and treatment, vitality and fatigue, physical mobility, pain and discomfort, sleep and rest, ability to work. Domain II: Mental domain: It covers body image and appearance, negative emotions, memory, and concentration. Domain III: Social domain: It covers the relationships with others, social support, and sexual life. Domain IV: Environmental domain: It covers financial resources, physical security, access to health services, home environment, opportunity for rest and recreation, physical environment and transportation. The quality of life increases as the score obtained from the domains increases .

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Başkaya, PhD, Principal Investigator — Uşak University Vocational School of Health Services 64000 Uşak / Turkey
Locations (1):
- Uşak Üniversity, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Other researchers will be able to read detailed information such as the research method and results when the research is published. The "Research Protocol" will be available on the this PRS page.